CLINICAL TRIAL: NCT06664931
Title: Muscle Energy Versus Mulligan Techniques in Treating Patients With Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Badier Elkomy, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005271
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cervical Spondylosis; Mulligan Mobilization; SNAGs; Muscle Energy Technique; Post Isometric Relaxation
Keywords: Mulligan Mobilization; Mobilization with Movement; SNAGs; Muscle Energy Technique; Post isometric relaxation; Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Population Groups; 2-methylcyclopentadienyl manganese tricarbonyl

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) Muscle Energy Technique (MET). (Experimental): These participants will receive METs, in addition to a standard physical therapy program consisting of deep neck flexor strengthening exercises, isometric exercise, and range of motion exercises (3 sessions per week for 4 weeks).
  Interventions: Other: Group (A) Muscle Energy Technique (MET)
- Group (B) Mulligan Mobilization Technique group (MMT). (Experimental): Participants will receive MMT interventions alongside the standard physical therapy program deep neck flexor strengthening exercises, isometric exercise, and range of motion exercises 3 sessions per week for 4 weeks.
  Interventions: Other: Group (B) Mulligan Mobilizations Techniques (MMT).

INTERVENTIONS:
Other: Group (A) Muscle Energy Technique (MET) — MET will be applied to three key muscles commonly associated with neck pain:
  upper trapezius, levator scapulae, and anterior scalenus.
  Other Names: Post Isometric Relaxation
  Arms: Group (A) Muscle Energy Technique (MET).
Other: Group (B) Mulligan Mobilizations Techniques (MMT). — Participants in Group (B) will receive MMT alongside the traditional treatment. MMT utilizes a specific technique called Sustained Natural Apophyseal Glides (SNAGs) to improve joint mobilization.
  Other Names: SNAGs
  Arms: Group (B) Mulligan Mobilization Technique group (MMT).

SUMMARY:
This study will be aimed to answer the following questions:

Which technique, MET or MMT, is more effective in reducing pain, increasing range of motion (ROM), improving proprioception, and enhancing functional ability in individuals with CS?

It will be assumed that:

1. All participants will adhere to study instructions and procedures.
2. All participants will be evaluated under standardized conditions.

DETAILED DESCRIPTION:
Cervical spondylosis (CS) is a highly prevalent age-related condition (95%), that affects the joints and discs of the cervical spine. By age 65, nearly all individuals experience some degree of degeneration, characterized by disc breakdown and enlarged facet joints. While aging is the primary cause, injuries can accelerate this process in younger populations.

Significance of the Study Age-related degenerative spinal changes are almost widespread. Population-based studies have shown that approximately 80 to 90% of people have disk degeneration on magnetic resonance imaging (MRI) by the age of 50 years.

A global burden review estimates that over 300 million people worldwide had mechanical neck pain lasting at least 3 months in 2015.

Clinical features of spondylosis are more common in men than in women, with a peak incidence between the ages of 40 and 60 years for both men and women.

Cervical spondylosis commonly affects the middle and lower cervical vertebrae (C5-C6 and C6-C7), although higher levels may also be involved. Neck pain is the most prominent symptom. CS can affect all cervical components (i.e., the spinal cord, spinal vasculature, and nerve roots). Cervical spondylosis Symptoms include cervical instability (abnormal movement or laxity between vertebrae). This instability can lead to various symptoms such as neck pain, muscle imbalance between cervical and shoulder girdle muscles (weakness in cervical flexors, lower trapezius, and anterior serratus; tightness in the upper trapezius, scapular lift, and pectoralis major), disc herniation and osteophyte formation. These can compromise proprioception (accurate sensory feedback) and limit neck mobility, significantly impacting function and daily activities.

Muscle energy techniques is a form of manual therapy frequently used by physical therapists to improve musculoskeletal function and alleviate pain. MET aims to adjust abnormal muscle tone by training specific muscles, enhancing strength and stability, improving the musculoskeletal function, and ultimately improving quality of life.

Another treatment technique is MMT that is now an integral component of many manual physiotherapists' clinical practice. MMT involves sustained passive accessory force/glide to a joint while the participant actively performs a problematic movement.

This study aims to address this gap in knowledge by investigating whether MET or MMT is more effective in improving pain, ROM, proprioception, and functional ability in individuals with cervical spondylosis. The findings from this study can provide valuable insights for physical therapists in selecting the most appropriate treatment approach for their patients with cervical spondylosis. By determining the more effective technique, physical therapists can optimize treatment plans and potentially improve patient outcomes.

This Triple-blinded (the examiner, statistician, and the participants will be blinded, while the therapist will be aware of treatment procedures) randomized controlled trial (RCT) will investigate the effectiveness of Muscle Energy Techniques (MET) compared to Mulligan Mobilization Techniques (MMT) on cervical spine pain, ROM, and function in participants with Cervical Spondylosis (CS). The study will be conducted at the outpatient physical therapy clinic of Horus University in New Damietta, Egypt.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of both genders aged 40 - 60 years old, diagnosed with clinically and medically stable CS.
2. All participants will be assessed and referred by orthopedic surgeons before starting the study.
3. Mechanical neck pain localized to the cervical.
4. Neck pain lasting more than 3 months, local tenderness of the upper fibers of the trapezius, limitation in cervical ROM and muscle spasm.
5. Moderate pain intensity (45-74 mm on VAS).
6. Participants with Moderate pain intensity NDI (30 - 48%).
7. All participants are free from any pathological conditions that might influence the results.

Exclusion Criteria:

1. Participants with systemic diseases like rheumatoid arthritis, metabolic diseases, or osteoporosis.
2. History of trauma or accidental injuries to the cervical spine.
3. Cervical myelopathy, inflammatory arthritis, tumors, infections involving the cervical spine, or vertebrobasilar artery insufficiency.
4. Cervical spine injury, dizziness, vertigo, or any other musculoskeletal complaints.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion (CROM) | Pre- intervention and after 4 weeks of treatment
  to measure the Cervical ROM for (Flexion, Extension, Rotation for both sides and Sidebending for both sides) and proprioception (Neutral head position test, and Target head position)
The Arabic Version Of Neck Disability Index (NDI). | Pre- intervention and after 4 weeks of treatment
  to assess the level of disabilities in patients with neck pain, in % points
Visual Analogue Scale (VAS). | Pre- intervention and after 4 weeks of treatment
  to measure neck pain with score extended from 0 to 10, minimum score 0 (no pain), highest score 10 (worst pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Horus University - Egypt, Cairo, Egypt

REFERENCES:
- [Background] Binch AL, Cole AA, Breakwell LM, Michael AL, Chiverton N, Creemers LB, Cross AK, Le Maitre CL. Nerves are more abundant than blood vessels in the degenerate human intervertebral disc. Arthritis Res Ther. 2015 Dec 21;17:370. doi: 10.1186/s13075-015-0889-6. PMID 26695177
- [Background] Manzoor A, Anwar N, Khalid K, Haider R, Saghir M, Javed MA. Comparison of effectiveness of muscle energy technique with Mulligan mobilization in patients with non-specific neck pain. J Pak Med Assoc. 2021 Jun;71(6):1532-1524. doi: 10.47391/JPMA.981. PMID 34111066
- [Background] Atisook R, Euasobhon P, Saengsanon A, Jensen MP. Validity and Utility of Four Pain Intensity Measures for Use in International Research. J Pain Res. 2021 Apr 21;14:1129-1139. doi: 10.2147/JPR.S303305. eCollection 2021. PMID 33907460
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Bagcaci S, Unuvar BS, Gercek H, Ugurlu I, Sert OA, Yilmaz K. A randomized controlled trial on pain, grip strength, and functionality in lateral elbow pain: Mulligan vs muscle energy techniques. J Back Musculoskelet Rehabil. 2023;36(2):419-427. doi: 10.3233/BMR-220061. PMID 36120766
- [Background] Bakhsheshian J, Mehta VA, Liu JC. Current Diagnosis and Management of Cervical Spondylotic Myelopathy. Global Spine J. 2017 Sep;7(6):572-586. doi: 10.1177/2192568217699208. Epub 2017 May 31. PMID 28894688
- [Background] Baron EM, Young WF. Cervical spondylotic myelopathy: a brief review of its pathophysiology, clinical course, and diagnosis. Neurosurgery. 2007 Jan;60(1 Supp1 1):S35-41. doi: 10.1227/01.NEU.0000215383.64386.82. PMID 17204884
- [Background] Binder AI. Cervical spondylosis and neck pain. BMJ. 2007 Mar 10;334(7592):527-31. doi: 10.1136/bmj.39127.608299.80. No abstract available. PMID 17347239
- [Background] Bono CM, Ghiselli G, Gilbert TJ, Kreiner DS, Reitman C, Summers JT, Baisden JL, Easa J, Fernand R, Lamer T, Matz PG, Mazanec DJ, Resnick DK, Shaffer WO, Sharma AK, Timmons RB, Toton JF; North American Spine Society. An evidence-based clinical guideline for the diagnosis and treatment of cervical radiculopathy from degenerative disorders. Spine J. 2011 Jan;11(1):64-72. doi: 10.1016/j.spinee.2010.10.023. PMID 21168100
- [Background] Brinjikji W, Luetmer PH, Comstock B, Bresnahan BW, Chen LE, Deyo RA, Halabi S, Turner JA, Avins AL, James K, Wald JT, Kallmes DF, Jarvik JG. Systematic literature review of imaging features of spinal degeneration in asymptomatic populations. AJNR Am J Neuroradiol. 2015 Apr;36(4):811-6. doi: 10.3174/ajnr.A4173. Epub 2014 Nov 27. PMID 25430861
- [Background] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800
- [Background] Cheung J, Kajaks T, Macdermid JC. The relationship between neck pain and physical activity. Open Orthop J. 2013 Sep 20;7:521-9. doi: 10.2174/1874325001307010521. eCollection 2013. PMID 24133553
- [Background] Copurgensli C, Gur G, Tunay VB. A comparison of the effects of Mulligan's mobilization and Kinesio taping on pain, range of motion, muscle strength, and neck disability in patients with Cervical Spondylosis: A randomized controlled study. J Back Musculoskelet Rehabil. 2017;30(1):51-62. doi: 10.3233/BMR-160713. PMID 27257980
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Dong WK, Lin XH. [Clinical observation on cervical spondylosis of neck type treated with acupuncture at original and terminal points of trapezius]. Zhongguo Zhen Jiu. 2012 Mar;32(3):211-4. Chinese. PMID 22471131
- [Background] van Eerd M, Patijn J, Loeffen D, van Kleef M, Wildberger J. The Diagnostic Value of an X-ray-based Scoring System for Degeneration of the Cervical Spine: A Reproducibility and Validation Study. Pain Pract. 2021 Sep;21(7):766-777. doi: 10.1111/papr.13013. Epub 2021 May 18. PMID 33837629
- [Background] Emery SE. Cervical spondylotic myelopathy: diagnosis and treatment. J Am Acad Orthop Surg. 2001 Nov-Dec;9(6):376-88. doi: 10.5435/00124635-200111000-00003. PMID 11767723
- [Background] Exelby L. The Mulligan concept: its application in the management of spinal conditions. Man Ther. 2002 May;7(2):64-70. doi: 10.1054/math.2001.0435. PMID 12374089
- [Background] Ferrara LA. The biomechanics of cervical spondylosis. Adv Orthop. 2012;2012:493605. doi: 10.1155/2012/493605. Epub 2012 Feb 1. PMID 22400120
- [Background] Franke H, Fryer G, Ostelo RW, Kamper SJ. Muscle energy technique for non-specific low-back pain. Cochrane Database Syst Rev. 2015 Feb 27;2015(2):CD009852. doi: 10.1002/14651858.CD009852.pub2. PMID 25723574
- [Background] Ghasemi M, Golabchi K, Mousavi SA, Asadi B, Rezvani M, Shaygannejad V, Salari M. The value of provocative tests in diagnosis of cervical radiculopathy. J Res Med Sci. 2013 Mar;18(Suppl 1):S35-8. PMID 23961282
- [Background] Gillani SN, Ain Q-, Rehman SU, Masood T. Effects of eccentric muscle energy technique versus static stretching exercises in the management of cervical dysfunction in upper cross syndrome: a randomized control trial. J Pak Med Assoc. 2020 Mar;70(3):394-398. doi: 10.5455/JPMA.300417. PMID 32207413
- [Background] Gugliotti M, Tau J, Gallo K, Sagliocca N, Horan M, Sussman N, Wisnewski R. Between-week reliability of the cervical range of motion (CROM) device for upper cervical rotation. J Man Manip Ther. 2021 Jun;29(3):176-180. doi: 10.1080/10669817.2020.1805691. Epub 2020 Aug 18. PMID 32808588
- [Background] Haladaj R, Pingot M, Topol M. The Effectiveness of Cervical Spondylosis Therapy with Saunders Traction Device and High-Intensity Laser Therapy: A Randomized Controlled Trial. Med Sci Monit. 2017 Jan 20;23:335-342. doi: 10.12659/msm.899454. PMID 28104903
- [Background] Hanks J, Myers B. Validity, Reliability, and Efficiency of a Standard Goniometer, Medical Inclinometer, and Builder's Inclinometer. Int J Sports Phys Ther. 2023 Aug 1;18(4):989-996. doi: 10.26603/001c.83944. eCollection 2023. PMID 37547826
- [Background] Hartley KG, Damon BM, Patterson GT, Long JH, Holt GE. MRI techniques: a review and update for the orthopaedic surgeon. J Am Acad Orthop Surg. 2012 Dec;20(12):775-87. doi: 10.5435/JAAOS-20-12-775. PMID 23203937
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] Hussien HM, Abdel-Raoof NA, Kattabei OM, Ahmed HH. Effect of Mulligan Concept Lumbar SNAG on Chronic Nonspecific Low Back Pain. J Chiropr Med. 2017 Jun;16(2):94-102. doi: 10.1016/j.jcm.2017.01.003. Epub 2017 Mar 30. PMID 28559749
- [Background] Jaiswal PR, Qureshi I, Phansopkar PA. Effectiveness of Mulligan's Two-Leg Rotation Versus Muscle Energy Technique in Subjects With Hamstring Tightness. Cureus. 2022 Sep 7;14(9):e28890. doi: 10.7759/cureus.28890. eCollection 2022 Sep. PMID 36225495
- [Background] Kashyap R, Iqbal A, Alghadir AH. Controlled intervention to compare the efficacies of manual pressure release and the muscle energy technique for treating mechanical neck pain due to upper trapezius trigger points. J Pain Res. 2018 Dec 12;11:3151-3160. doi: 10.2147/JPR.S172711. eCollection 2018. PMID 30588067
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187
- [Background] Ptaszkowski K, Slupska L, Paprocka-Borowicz M, Kolcz-Trzesicka A, Zwierzchowski K, Halska U, Przestrzelska M, Mucha D, Rosinczuk J. Comparison of the Short-Term Outcomes after Postisometric Muscle Relaxation or Kinesio Taping Application for Normalization of the Upper Trapezius Muscle Tone and the Pain Relief: A Preliminary Study. Evid Based Complement Alternat Med. 2015;2015:721938. doi: 10.1155/2015/721938. Epub 2015 Aug 12. PMID 26347792
- [Background] Pumberger M, Froemel D, Aichmair A, Hughes AP, Sama AA, Cammisa FP, Girardi FP. Clinical predictors of surgical outcome in cervical spondylotic myelopathy: an analysis of 248 patients. Bone Joint J. 2013 Jul;95-B(7):966-71. doi: 10.1302/0301-620X.95B7.31363. PMID 23814251
- [Background] Razzaq A, Nadeem RD, Akhtar M, Ghazanfar M, Aslam N, Nawaz S. Comparing the effects of muscle energy technique and mulligan mobilization with movements on pain, range of motion, and disability in adhesive capsulitis. J Pak Med Assoc. 2022 Jan;72(1):13-16. doi: 10.47391/JPMA.1360. PMID 35099430
- [Background] Reddy RS, Tedla JS, Dixit S, Abohashrh M. Cervical proprioception and its relationship with neck pain intensity in subjects with cervical spondylosis. BMC Musculoskelet Disord. 2019 Oct 15;20(1):447. doi: 10.1186/s12891-019-2846-z. PMID 31615495
- [Background] Reyhan AC, Sindel D, Dereli EE. The effects of Mulligan's mobilization with movement technique in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2020;33(1):99-107. doi: 10.3233/BMR-181135. PMID 31104005
- [Background] Rostron S. The Effects of Massage Therapy on a Patient with Migraines and Cervical Spondylosis: a Case Report. Int J Ther Massage Bodywork. 2021 Sep 2;14(3):15-21. doi: 10.3822/ijtmb.v14i3.629. eCollection 2021 Sep. PMID 34484491
- [Background] Ahmed A, Ibrar M, Arsh A, Wali S, Hayat S, Abass S. Comparing the effectiveness of Mulligan mobilization versus Cyriax approach in the management of patients with subacute lateral epicondylitis. J Pak Med Assoc. 2021 Jan;71(1(A)):12-15. doi: 10.47391/JPMA.186. PMID 33484510
- [Background] Rubinstein SM, Pool JJ, van Tulder MW, Riphagen II, de Vet HC. A systematic review of the diagnostic accuracy of provocative tests of the neck for diagnosing cervical radiculopathy. Eur Spine J. 2007 Mar;16(3):307-19. doi: 10.1007/s00586-006-0225-6. Epub 2006 Sep 30. PMID 17013656
- [Background] Sadeghi A, Rostami M, Ameri S, Karimi Moghaddam A, Karimi Moghaddam Z, Zeraatchi A. Effectiveness of isometric exercises on disability and pain of cervical spondylosis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Jun 16;14(1):108. doi: 10.1186/s13102-022-00500-7. PMID 35710510
- [Background] Sbardella S, La Russa C, Bernetti A, Mangone M, Guarnera A, Pezzi L, Paoloni M, Agostini F, Santilli V, Saggini R, Paolucci T. Muscle Energy Technique in the Rehabilitative Treatment for Acute and Chronic Non-Specific Neck Pain: A Systematic Review. Healthcare (Basel). 2021 Jun 17;9(6):746. doi: 10.3390/healthcare9060746. PMID 34204590
- [Background] Shaheen AA, Omar MT, Vernon H. Cross-cultural adaptation, reliability, and validity of the Arabic version of neck disability index in patients with neck pain. Spine (Phila Pa 1976). 2013 May 1;38(10):E609-15. doi: 10.1097/BRS.0b013e31828b2d09. PMID 23429690
- [Background] Shedid D, Benzel EC. Cervical spondylosis anatomy: pathophysiology and biomechanics. Neurosurgery. 2007 Jan;60(1 Supp1 1):S7-13. doi: 10.1227/01.NEU.0000215430.86569.C4. PMID 17204889
- [Background] Smith M, Fryer G. A comparison of two muscle energy techniques for increasing flexibility of the hamstring muscle group. J Bodyw Mov Ther. 2008 Oct;12(4):312-7. doi: 10.1016/j.jbmt.2008.06.011. Epub 2008 Aug 6. PMID 19083689
- [Background] Steilen D, Hauser R, Woldin B, Sawyer S. Chronic neck pain: making the connection between capsular ligament laxity and cervical instability. Open Orthop J. 2014 Oct 1;8:326-45. doi: 10.2174/1874325001408010326. eCollection 2014. PMID 25328557
- [Background] Takagi I, Eliyas JK, Stadlan N. Cervical spondylosis: an update on pathophysiology, clinical manifestation, and management strategies. Dis Mon. 2011 Oct;57(10):583-91. doi: 10.1016/j.disamonth.2011.08.024. No abstract available. PMID 22036114
- [Background] Theodore N. Degenerative Cervical Spondylosis. N Engl J Med. 2020 Jul 9;383(2):159-168. doi: 10.1056/NEJMra2003558. No abstract available. PMID 32640134
- [Background] Tu J, Vargas Castillo J, Das A, Diwan AD. Degenerative Cervical Myelopathy: Insights into Its Pathobiology and Molecular Mechanisms. J Clin Med. 2021 Mar 15;10(6):1214. doi: 10.3390/jcm10061214. PMID 33804008
- [Background] Thomas E, Cavallaro AR, Mani D, Bianco A, Palma A. The efficacy of muscle energy techniques in symptomatic and asymptomatic subjects: a systematic review. Chiropr Man Therap. 2019 Aug 27;27:35. doi: 10.1186/s12998-019-0258-7. eCollection 2019. PMID 31462989
- [Background] Uysal SC, Tuzun EH, Eker L, Angin E. Effectiveness of the muscle energy technique on respiratory muscle strength and endurance in patients with fibromyalgia. J Back Musculoskelet Rehabil. 2019;32(3):411-419. doi: 10.3233/BMR-181287. PMID 30475751
- [Background] Venosa M, Romanini E, Padua R, Cerciello S. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation in patients with cervical spondylosis: a randomized controlled trial. Lasers Med Sci. 2019 Jul;34(5):947-953. doi: 10.1007/s10103-018-2682-7. Epub 2018 Nov 15. PMID 30443883
- [Background] Xiong J, Zhang Z, Zhang Z, Ma Y, Li Z, Chen Y, Liu Q, Liao W. Short-term effects of Kinesio taping combined with cervical muscles multi-angle isometric training in patients with cervical spondylosis. BMC Musculoskelet Disord. 2023 Jan 18;24(1):38. doi: 10.1186/s12891-023-06154-x. PMID 36650475
- [Background] Yang J, Lee B, Kim C. Changes in proprioception and pain in patients with neck pain after upper thoracic manipulation. J Phys Ther Sci. 2015 Mar;27(3):795-8. doi: 10.1589/jpts.27.795. Epub 2015 Mar 31. PMID 25931733
- [Background] Young IA, Michener LA, Cleland JA, Aguilera AJ, Snyder AR. Manual therapy, exercise, and traction for patients with cervical radiculopathy: a randomized clinical trial. Phys Ther. 2009 Jul;89(7):632-42. doi: 10.2522/ptj.20080283. Epub 2009 May 21. PMID 19465371
- [Background] Zaidi F, Ahmed I. Effectiveness of muscle energy technique as compared to Maitland mobilisation for the treatment of chronic sacroiliac joint dysfunction. J Pak Med Assoc. 2020 Oct;70(10):1693-1697. doi: 10.5455/JPMA.43722. PMID 33159735